CLINICAL TRIAL: NCT05722535
Title: Using Shared Decision Making to Improve Family Media Use Planning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Kroshus, Research Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R21HD107230 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Behavior
Keywords: Screen Media Use
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed FMC (No Intervention): Families assigned to the control condition will receive the FMC after study completion.
- FMC (Experimental): Families randomized to the intervention condition will receive the FMC after they complete the baseline survey.
  Interventions: Behavioral: Family Media Check-In (FMC)

INTERVENTIONS:
Behavioral: Family Media Check-In (FMC) — An interactive, web-based tool to support within-family media use planning will be developed and shared with families.
  Arms: FMC

SUMMARY:
Investigators will conduct a pilot randomized controlled trial assessing the efficacy and feasibility of the newly developed Family Media Check-In (FMC).

DETAILED DESCRIPTION:
The clinical trial portion of this study will enroll 150 families (child age 11-17, and at least one parent/guardian). Stratified randomization will be used to assign families to the intervention (FMC) or control (delayed FMC) condition. Families assigned to the intervention condition will be asked to complete the FMC within 2 weeks of randomization and will be sent a second survey one week after completion. Participants in the control condition will complete a condition-specific subset of these questions three weeks after baseline. Participants in both conditions will complete a follow-up survey two months after their second survey.

The primary outcomes will be measured at the first follow-up period and will be related to screen media planning and decision making. Two-month follow-up surveys will explore intervention impact on screen media practices.

Prior to the clinical trial portion of the study, the study team conducted interviews/focus groups, participatory design sessions, and usability testing sessions with a diverse group of families to refine the concept for the intervention and to iteratively develop the intervention itself. Changes in the behavioral targets and components of the intervention and outcomes for the evaluation (relative to the original grant proposal) were driven by family-expressed needs and priorities.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 11 and 17
* Parent/guardian of a child between the ages of 11 and 17
* English speaking

Exclusion Criteria:

* Parent/guardian or child does not want to participate (i.e., dyads only)
* Non-English speaking

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Decision Satisfaction | Baseline, 3 weeks post-baseline
  Perceived Effective Decision Scale: a 4-item measure that assesses parent and teen satisfaction with their family media plan. Responses are measured on a 5-point Likert scale, with higher scores indicating a stronger perception of decision effectiveness.
Decision Uncertainty | Baseline, 3 weeks post-baseline
  Decision Uncertainty Scale: a 3-item scale adapted for the intervention and nature of decision designed to measure parent and teen perceptions of uncertainty when making decisions. The items evaluate factors contributing to uncertainty, including difficulty, lack of clarity, and indecision. Responses are recorded on a 5-point Likert scale. Higher scores indicate greater levels of perceived uncertainty, with the third item reverse-scored.
Change in Family Media Planning and Plan Engagement | Baseline, 3 weeks post-baseline
  Family Media Planning and Engagement Scale. This scale includes two components, each with 3 items: elements included in plan and engagement with plan. Higher scores indicate more screen media-related elements included in plan and greater teen engagement with plan.
Teen Involvement in Plan | Baseline, 3 weeks post-baseline
  This single-item assesses the degree of involvement teens perceive they had in creating the plan. Response options range from full individual control to full parent parental control, with options capturing varying levels of shared-decision making

SECONDARY OUTCOMES:
Screen Media Conflict | Baseline, 3 weeks post-baseline
  3 items from the 2003 PEW Research Center Survey about how often parents and teens have argued in the past 2 weeks about three dimensions of teen screen media use.
Screen-Related Parenting Style | Baseline, 3 weeks post-baseline
  Perceived Parental Media Mediation Scale: a 15-item measure adapted for the main types of digital media use addressed in the intervention that assess teen perceptions of restrictive and active parental mediation. Responses are recorded on a 5-point Likert scale; responses to items are added together to create a total score, with higher scores indicating a greater perception of parental media mediation.
Acceptability of FMC | 1 week post-intervention / 3 weeks post-baseline
  Acceptability of Intervention Measure: a 4 item 4 point Likert scale with higher score indicating a higher level of acceptability

OTHER OUTCOMES:
Amount of Use | Baseline, 3 weeks post-baseline
  Parent and teen self-report of screen media use during a typical weekday and weekend for something other than school or work. Response options range from "I did not use screen media" to "6 or more hours".
Social Media Addiction | Baseline, 3 weeks post-baseline
  Bergen Social Media Addiction Scale: a 6-item measure to assess teen-reported dependence on social media. Each of the 6 items are rated on a 5-point Likert scale, with higher scores indicating a greater risk of social media addiction.
Change in Problematic Media use | Baseline, 3 weeks post-baseline
  Problematic Media Use Measure - Short Form: a 9-item scale which measures elements of addictive media use among children, including preoccupation, withdrawal, and unsuccessful attempts to control use by parents. Responses are recorded on a 5 point Likert scale with higher scores indicating more problematic media use.
Parent Distracted Media Use | Baseline, 3 weeks post-baseline
  Parent self-report and teen report of parent behavior. A single item question that measures how frequently parents are perceived as being distracted by their smartphones during conversations with their children. It is assessed using a question adapted from a PEW Center questionnaire, asked to both parents and teens. Response options include: often, sometimes, rarely, never distracted, or I/my parent does not have a smartphone.
Emotional Health | Baseline, 3 weeks post-baseline
  PedsQL Emotional Health subscale: A 5-item measure that assess emotional health in adolescents, focusing on the frequency of emotions such as sadness, anger, worry, or difficulty sleeping. ) Responses are recorded on a 5-point Likert scale (1=not at all to 5=very much), with higher scores reflecting higher levels of emotional well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No